CLINICAL TRIAL: NCT06664034
Title: Intervening on Women's Health for Rural Young Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: San Diego State University (Other); Cancer Resource Center of the Desert (Unknown); El Centro Regional Medical Center (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Hui-Chun Irene Su, Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: U54800646; 5U54CA285115-02 (NIH)
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Cancer; Fertility Issues; Contraception
Keywords: Reproductive health; Oncofertility
MeSH Terms: conditions — Neoplasms; Infertility

STUDY DESIGN:
Intervention Model Description: single arm pilot hybrid type I trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multi-component intervention (Experimental): After the intervention implementation, all cancer patients presenting to oncology clinical visits that meet eligibility criteria will receive the multi-component intervention.
  Interventions: Behavioral: Multi-component reproductive health care intervention

INTERVENTIONS:
Behavioral: Multi-component reproductive health care intervention — The multi-component reproductive health care intervention includes:
  1. Young cancer patients presenting to oncology visits will complete a clinic-based reproductive health needs screen with a member of the clinical team. This needs screen assesses i) desire to have a child in the future and ii) need for contraception.
  2. Reproductive health patient navigation consists of one telehealth or in-person session with a social worker to: i) assess the patient's reproductive health needs, ii) provide individualized patient education and counseling on a) infertility risk related to cancer type and treatment and b) screening and management strategies for reproductive health needs, iii) provide support with the goal of engaging in goal-concordant reproductive health care.
  3. Telehealth reproductive health consultation will occur between the patient and reproductive specialist. Each consultation is estimated to be 1 hour.

SUMMARY:
The purpose of this pilot study is to evaluate the feasibility of a multi-component intervention to improve young female cancer survivors' engagement in goal-concordant reproductive health care. The investigators hypothesize that implementation of the intervention will result in increased young cancer survivors' engagement in goal-concordant reproductive health care.

ELIGIBILITY:
Inclusion Criteria:

* Cancer (Stages 0-IV) diagnosis
* Primary language English or Spanish
* Receiving oncology care at rural oncology clinical participating site
* Living in Imperial County, California

Exclusion Criteria:

- Women who are pregnant at recruitment

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 64 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patient's engagement in goal-concordant reproductive health care | 12 weeks after oncology visit
  Study staff will be trained to abstract the primary outcome from the patient's medical records using standardized case report forms. Engagement in goal-concordant reproductive health care will be assigned to patients who undergo: 1) reproductive health needs screen and have no needs, OR 2) reproductive health needs screen, complete a navigation session and receive reproductive health counseling and management strategies, and have no further needs; OR 3) reproductive health needs screen, complete a navigation session and receive reproductive health counseling and management strategies, have a need, undergo a telehealth reproductive health consultation, and have no reproductive health service needs; OR 4) reproductive health needs screen, complete a navigation session and receive reproductive health counseling and management strategies, have a need, undergo a telehealth reproductive health consultation, have a reproductive health service needs, and uptake appropriate services.

CONTACTS AND LOCATIONS:
Overall Officials: H. Irene Su, MD, MSCE, Principal Investigator — University of California, San Diego
Locations (4):
- United States (4):
  - San Diego State University - Imperial Valley/ School of Nursing, Brawley, California
  - Cancer Resource Center of the Desert, El Centro, California
  - El Centro Regional Medical Center, El Centro, California
  - University of Califiornia San Diego, La Jolla, California

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data generated during the study will be available from the principal investigator (H. Irene Su) upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication.
Access Criteria: Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to the principal investigator (H. Irene Su).